CLINICAL TRIAL: NCT07367061
Title: Clinical Investigation to Assess Safety and Efficacy of INNEA AQUA in Adult Women With Vulvo-Vaginal Atrophy (VVA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innate srl (Industry)
Collaborators: CEBIS International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INN-AQA-10/24
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Vulvo Vaginal Atrophy
Keywords: VVA; hyaluronic acid; vulvo vaginal atrophy; vaginal atrophy

STUDY DESIGN:
Intervention Model Description: This is an open, double-arm, prospective, multicenter clinical investigation to evaluate the safety and efficacy of INNEA AQUA in adult women aged 18-75 with Vulvo-vaginal atrophy (VVA). The enrollment period will be 6 months, and the clinical investigation period will be up to 12 weeks per patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: randomized to the treatment Innea Aqua (Experimental): 31 women (18-75) treated with product Innea Aqua. 1 injection of the product and after 30 days another injection
  Interventions: Device: product: Innea Aqua vaginal use
- Arm 2: randomized to the treatment to the standard of care (Active Comparator): standard of care tratment
  Interventions: Device: arm 2: standard of care

INTERVENTIONS:
Device: product: Innea Aqua vaginal use — product object of the investigation: Innea Aqua for vaginal use, 2 mL product. Labelled as Innea Aqua.
  Arms: Arm 1: randomized to the treatment Innea Aqua
Device: arm 2: standard of care — the comparator is the standard of care selected by the centre
  Arms: Arm 2: randomized to the treatment to the standard of care

SUMMARY:
Clinical investigation to assess safety and efficacy of INNEA AQUA in adult women with Vulvo-Vaginal Atrophy (VVA).

To assess the Safety and efficacy of INNEA AQUA

DETAILED DESCRIPTION:
Clinical investigation to assess safety and efficacy of INNEA AQUA in adult women with Vulvo-Vaginal Atrophy (VVA).

To assess the Safety and efficacy of INNEA AQUA

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 18-75 (both fertile and post-menopausal)
* Vulvovaginal atrophy diagnostic
* Signed written informed consent.
* Vaginal Ph more than 4.5
* Willing to sign the informed consent form
* Willing to comply with the clinical investigation visits.

Exclusion Criteria:

* patients who tend to develop hypertrophic scarring,
* patients with a history of autoimmune disease or who are receiving immune therapy,
* patients who are known to be hypersensitive or allergic to hyaluronic acid and other INNEA AQUA components,
* pregnant or breastfeeding women,
* patients under 18 years of age,
* vagina with hypertrophic scars from different etiology,
* patients with presence of ≥ stage 2 apical pelvic organ prolapse,
* patients with stress urinary incontinence,
* patients with vaginismus, vulvovaginal or urinary tract infection,
* patients with Hemorrhagic or neoplastic genital pathologies or hormone-dependent tumor
* patients with genital bleeding of unknown etiology, recurrent porphyria, uncontrolled epilepsy, heart conduction disorders, recurrent angina, rheumatic fever, previous vulvovaginal or uro-gynecological surgery, and hemostatic disorders,
* Anticoagulated patients or patients receiving platelet aggregation inhibitors should not be treated with INNEA AQUA,
* INNEA AQUA must not be used in areas presenting inflammatory and/or infectious processes (e.g., papilloma, herpes). INNEA AQUA must not be used in association with other invasive treatments,
* Avoid using in combination with any other concomitant therapies for same indication;
* Patients who are using substances that can prolong bleeding (such as aspirin, nonsteroidal anti-inflammatory drugs, and warfarin) may, as with any injection, experience increased bruising or bleeding at treatment sites.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female (18-75 Years old)
Enrollment: 62 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
safety: Incidence of AE and SAE | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  To evaluate the safety of INNEA AQUA in adult participants. Incidence of adverse events, early withdrawal rate due to AEs, and device deficiencies, whether serious or not

SECONDARY OUTCOMES:
Efficacy: change in pruritus | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Pruritus (0-10 visual analogue scales (VAS)) on Day 0, Day 30, Day 51, and Day 120
Efficacy: Change in soreness | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Soreness (0-10 visual analogue scales (VAS)) on Day 0, Day 30, Day 51, and Day 120
Efficacy: change in dyspareunia | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Dyspareunia (0-10 visual analogue scales (VAS)) on Day 0, Day 30, Day 51, and Day 120
efficacy: change in irritation | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Irritation (0-10 visual analogue scales (VAS)) on Day 0, Day 30, Day 51, and Day 120
efficacy: evaluation of pH | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Vaginal Ph Normalization
efficacy: change in vaginal moisture | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Vaginal moisture - Modified Schirmer test (mm) change on Day 30, Day 51, and Day 120 compared with baseline
efficacy: change in VHX | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Vaginal Health Index (VHI) score on Day 30, Day 51, and Day 120
efficacy: evaluation of vaginal aging | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in Day-to-Day Impact of Vaginal Aging Questionnaire on Day 30, Day 51, and Day 120
safety (AE/SAE) | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Incidence of adverse events, early withdrawal rate due to AEs, and device deficiencies, whether serious or not
efficacy: satisfaction of the patient | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Participant satisfaction in using the Device (PGI-I) Day 120
efficacy: satisfaction of the investigator | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Investigator satisfaction in using the Device (VAS) Day 120
efficacy: evaluation of quality of life | From enrollment to the end of treatment and second follow up visit at 120 days from the first injection
  Change in baseline score in QoL score when compared to Day 30, 51 and 120.

CONTACTS AND LOCATIONS:
Locations (3):
- Romania (3):
  - Obstretics and Gynaecology Filantropia Clinical Hospital, Bucharest, Romania
  - Nicolae Malaxa Clinical Hospital, Bucharest, Romania
  - AMCA Medical Clinic, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No